CLINICAL TRIAL: NCT04261803
Title: Familial Hypercholesterolemia Non Invasive Detection in Children by Salivary Test
Brief Title: FH Detection in Children by Salivary Test
Acronym: DEPEDIACOL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0861; 2019-A03076-51 (Other: ID-RCB)
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Hyperlipoproteinemia Type II
Keywords: familial hypercholesterolemia; Healthy Volunteers
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva and blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Familial Hypercholesterolemia children
  Interventions: Biological: salivary sample; Biological: blood test
- Control children
  Interventions: Biological: salivary sample; Biological: blood test

INTERVENTIONS:
Biological: salivary sample — spit of saliva in a tube
Biological: blood test — 2millilitter blood test

SUMMARY:
Familial Hypercholesterolemia is a common cause of premature coronary heart disease, it is present in 1 per 500 to 1 per 250 people of the general population. Studies on families of Hypercholesterolemia have shown that children with Hypercholesterolemia have a major increase in risk of coronary heart disease after the age of 20. The difference between Hypercholesterolemia and normal children in their atherogenic profil begin at the age of Nowadays , systematic screening techniques are not well implemented whereas their are clear World health organization guidelines.

International studies show treatment must be initiated early as at the age of eight years old.

In pediatry, Parents can be reluctant to practice blood test on their children. In order to allow more patients to be diagnosed and treated early enough to prevent major complications we need to find an non invasive test.

The main objective is to define the level of detection of cholesterol in saliva with two enzymatic tests. Furthermore we aim to evaluate the performance of salivary detection of cholesterol in children.

ELIGIBILITY:
Inclusion Criteria :

* children under 18 years old, with familial hypercholesterolemia
* children under 18 years old, intending surgery
* being able to spit

Exclusion Criteria:

* poor dental health
* for control patients: to have a known cholesterol disease

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Familial Hypercholesterolemia children group Control children group
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
salivary cholesterol concentration | Day 1
  the sample will be obtained during one visit non dedicated to this study (following-visit in nutrition for hypercholesterolemia children and before surgery for control children), the swabs of all the 60 patients will be used in two different methods of enzymatic tests.

CONTACTS AND LOCATIONS:
Overall Officials: Noel PERETTI, MD, Principal Investigator — Hospices Civils de Lyon gastro-enterological hepatology and nutrition
Locations (1):
- Hospices Civils de Lyon gastro-enterological hepatology and nutrition, Bron, France